CLINICAL TRIAL: NCT03279445
Title: Characteristics of African American People With Parkinson's Disease: A Hospital Based Study at the University of Chicago of the African American Community in Chicago's South Side
Brief Title: Parkinson's Disease in African American and Caucasian Patients
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 17-0998
Record Dates: First submitted 2017-08-14; First posted 2017-09-12 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — As described in the Study Description above for details on study design. Two tubes of blood of 8 ml each will be obtained from patients for future genetic testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- African American: Patient of African American race
- Caucasian: Patient of Caucasian race

SUMMARY:
More than 10 million people worldwide are living with Parkinson's disease (PD). While the actual number of African American (or Black) patients with PD is unknown, it is clear that there are racial disparities in the access to health care, diagnosis, treatment and survival of PD. The lack of clear knowledge on the possibly lower PD prevalence among African Americans compared to Caucasians further calls for more research in this field. The University of Chicago Medicine is an ideal facility to study this topic, due to its location on the South Side of Chicago with a large African American (or Black) population. By analyzing the demographics, socioeconomics and clinical features of PD patients in our Center for Research Informatics in African American (or Black) patients compared to the Caucasians of similar geographical area, the investigators aim to work toward a better understanding of the unique features of PD in American American (or Black) population, which might help improve the healthcare among this population in the Chicago and possibly nationwide as well.

DETAILED DESCRIPTION:
The first portion of the study will be a large medical electronic data based search and analysis of patients with PD on demographics, socioeconomic status and clinical features of PD patients. Specifically, we will retrospectively identify PD patients on both races from the electronic medical database spanned from 1/1/2006 to 10/31/2017 and compared demographics, socioeconomic status (educations, incomes and insurances), co-morbidities (all categories, including mood, cognition and psychosis), treatment (medications for parkinsonism and major non-motor symptoms, and frequency and locations of healthcare) and survival, and identified factors associated with medication usage and survival.

The second portion was designed to collect more detailed clinical assessments for information not available in the database and blood draws for genetic or candidate gene mutation analysis. Unfortunately, this part of the study could not be carried out due to the COVID-19 pandemic, which began shortly after completion of the first portion of the study. These assessments and analyses would have helped determine if there are significant differences in the clinical and genetic profiles between the African American (or Black) and Caucasian PD patients that account for their differences in clinical features and PD prevalence in these two populations.

ELIGIBILITY:
Inclusion Criteria:

* 15 years and older, confirmed diagnosis of PD, African American (or Black) or Caucasian race

Exclusion Criteria: Non-PD

-

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parkinson's patients of either African American (or Black) or Caucasian race.
Sampling Method: Non-Probability Sample
Enrollment: 2033 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Disparities in diagnosis, treatment and survival between Black and White Parkinson patients | Through study completion, an average of one year
  We will compare Black/AA and White PD patients on demographics, socioeconomic status (education, income, and insurance), co-morbidities, treatment (medications for parkinsonism and major non-motor symptoms, and frequency and locations of healthcare) and survival, and identify factors associated with medication usage and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Xie, MD, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xie T, Liao C, Lee D, Yu H, Padmanaban M, Kang W, Johnson J, Alshaikh J, Yuen C, Burns M, Chiu BC. Disparities in diagnosis, treatment and survival between Black and White Parkinson patients. Parkinsonism Relat Disord. 2021 Jun;87:7-12. doi: 10.1016/j.parkreldis.2021.04.013. Epub 2021 Apr 21. PMID 33905958